CLINICAL TRIAL: NCT05293379
Title: Prospective, Multicenter Study Assessing a Screening Campaign for Cardiovascular Diseases Risk Factors During SARS-CoV-2 Epidemic
Acronym: VACCIPREV
Status: Completed | Type: Observational
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: VACCIPREV
Record Dates: First submitted 2022-03-11; First posted 2022-03-24 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Health Behavior; Cardiovascular Diseases; Cardiovascular Morbidity
Keywords: cardiovascular risk factors; public health; screening campaign; cardiovascular disease; prevention; medical management
MeSH Terms: conditions — Health Behavior; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients sensitized in the VACCIPREV program: Patients from 3 vaccination centers who agreed to participate to the VACCIPREV program by using the teleconsultation booth and completing the questionnaires of tobacco dependance and assessment of sleep quality.
  Interventions: Other: Connected teleconsultation booth

INTERVENTIONS:
Other: Connected teleconsultation booth — 15-minutes assessment in a connected teleconsultation booth.

SUMMARY:
The goal of this prospective study is to evaluate the impact of an innovative screening campagn (using the medical device "CONSULT STATION®" on french population healthcare . The main aims of this study are:

* To determine whether a screening campaign for cardiovascular disease risk factor has a greater impact on the population who is not monitored by a primary care physician
* To determine whether people who are not monitored by a primary care physician have greater cardiovascular risk
* To determine whether the screening campaign offered to the general population has strengthened the relationship between community medecine and healthcare circuit coordination

Data of patients from vaccination center who agreed to participate to the screening campaign by using the medical device "CONSULT STATION®" will be analyzed.

Patients will also be called at least 3 months after their visit in the vaccination center in order to assess the impact of the screening campaign on their medical monitoring

DETAILED DESCRIPTION:
Cardiovascular diseases and its complications are the leading cause of death in the world. In France, they are the second leading cause of death after cancer, with over 140,000 deaths each year.

The number of people with cardiovascular disease increases with the aging of the population, and strong social and territorial inequalities persist. Innovative cardiovascular risk factors screening campaign can have significant public interest, especially to raise awareness and diagnose a particular population which is not monitored by a physician on a regular basis.

The VACCIPREV project emerged during the Covid-19 pandemic. The founding idea was to use the time people spent in vaccination centers to raise awareness and to diagnose people, for some, never go to a health facility. Indeed, a portion of the population free of all medical conditions, of all ages, including young people without known comorbidities, then crossed the threshold of our institutions to get vaccinated.

VACCIPREV is part of a global territorial prevention will to propose to this population flow an innovative medical technology optimizing all stages of vaccination.

In association with a French company named "H4D", developing a connected teleconsultation booth (CONSULT STATION®), an independent health check was thus structured, in addition with two questionnaires given during the waiting phase before vaccination: one concerning tobacco dependance and the other assessing the sleep quality. This health check focuses on the early detection of cardiovascular risk factors. It is indeed a key issue for medical management and VACCIPREV allows to respond to this issue in an innovative and playful way.

The CONSULT STATION® (Class IIa medical device certified according to European Directive 93/42/EEC) offers 15-minutes assessment of blood pressure, heart rate, oxygen saturation, BMI, but also the performance of visual tests. Accompanied by a caregiver in the process, the person gets in real time these different medical constants and thanks to a simple and graduated evaluation scale, a review of his results and a recommendation to visit his doctor if necessary. In case of potentially pathological results, and with the person's consent, contact informations (telephone/email) were collected to remotely assess the impact of this screening campaign.

VACCIPREV programme included an idependant medical check-up with the connected booth H4D, questionnaires of tabacco dependance and assessment of sleep quality and a remote assessment of their impact on the medical management of people with pathological constants. A telephone interview was carried out after a period of at least 3 months following the passage in the cabin to complete the medical questionnaire in order to evaluate changes in patients medical management. This included assessing the impact of the approach.

It was an observational study on data from an historic and prospective cohorte, multicentered national and not randomized. The study period was between 1st july 2021 and 1st july 2022.

The main objective of the study was to determine whether the innovative screening campaign has impacted the health management of the population.

Secondary objectives were:

* To determine whether the screening campaign's impact was greater in the population who is not monitored by a primary care physician
* To determine whether people who are not monitored by a physician have greater cardiovascular risk
* To determine whether the screening campaign offered to the general population has strengthened the relationship between community medecine and healthcare circuit coordination The objectives will be analysed both for all centers but aslo for each center in order to highlight a possible regional differences in the medical management of the population. Evaluation criteria concerning the objectives covered by this protocol will be based on a description of the data collected from the telephone interview (consultation with a general physician, consultation with a specialist, statement from a primary care physician)

ELIGIBILITY:
Inclusion Criteria:

* Patients informed of the study (information sheet given to patients) and who had not given their opposition to the collection of data for research purposes
* Woman or man aged 18 or over
* Patients registered with a social security scheme

Exclusion Criteria:

* Patients unable to understand the directives requested for the use of the cabin
* Patients under legal protection
* Patients who have expressed their opposition to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The targeting of patients covered the period from July 2021 to September 2021 corresponding to the period where the booth were available in vaccination centers. Data's extraction will extend from July 2021 to July 2022 in order to have a follow-up of at least 3 months after the passage in the cabin and to observe the potential modifications or initiation of patient care management.
  More than 6,000 people were sensitized within the framework of the VACCIPREV program, among them, about 2,400 patients have agreed to benefit from the independent assessment via the CONSULT STATION® within this same program in 3 months on the 3 sites. About 750 patients had a result with pathological constants and were invited to consult their attending physician.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of patients with pathological constants and have initiated a medical management | An average of 3 months
  Number of patients with pathological vitals and have initiated a medical management by a primary care physician or a specialist and whose constants'pathological criteria is confirmed by a physician

SECONDARY OUTCOMES:
Impact of the screening campaign in the population without a primary care physician | An average of 3 months
  Number of patients without a primary care physician with pathological findings and have initiated medical management by a general physician or a specialist and whose constant's pathological criteria is confirmed by the physician
Cardiovascular risk factors in the population without a primary care physician | An average of 3 months
  Comparison of cardiovascular disease risk factors in patients monitored by a primary care physician with patients who are not monitored by a primary care physician
Impact of the VACCIPREV program in strengthening the relationship between the community medecine and the coordination of healthcare circuits. | An average of 3 months
  The reinforcement of patients' reffering to community medecine will be evaluated with NECTAR software (establishment of the connection with community medicine)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Clinique de Saint Omer, Blendecques
  - Hôpital Privé Saint Claude, Saint-Quentin
  - Clinique Vauban, Valenciennes
  - Hôpital privé du Hainaut, Valenciennes

IPD SHARING:
Plan to Share IPD: No